CLINICAL TRIAL: NCT05023291
Title: Peroperative Assessment of Tumour Resection Margins Using High-resolution 18F-FDG-PET/CT in Pancreatic Adenocarcinoma, a Pilot Study: IMA PancreasCA (BC-05923)
Brief Title: Peroperative Assessment of Tumour Resection Margins Using High-resolution 18F-FDG-PET/CT in Pancreatic Adenocarcinoma
Acronym: IMA-PANC-CA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no effective result after first 5 patients
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BC-05923
Record Dates: First submitted 2020-08-24; First posted 2021-08-26 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- test group (Other): All patients who give their consent for this study will participate in the test group and will therefore receive the injection with 18F-FDG and images (PET / CT) will be made of the resection piece.
  Interventions: Diagnostic Test: Positron Emissie Tomografie - Computer Tomografie

INTERVENTIONS:
Diagnostic Test: Positron Emissie Tomografie - Computer Tomografie — In this study, the high-resolution PET-CT system will be used to evaluate the cutting edges after tumor resection. The goal is to evaluate the distance of the tumor cells from the cutting edges of the surgical piece. The patient receives an intravenous injection of radiolabeled sugar (18F-FDG). 18F-FDG is the standard PET tracer for diagnostic PET-CT research. This standard dose will always be calculated according to the formula: 3.7 x body weight + 37 Mbq.

SUMMARY:
One of the main risks for recurrence in patients with pancreatic cancer is incomplete surgery of the primary tumor. During the operation, the surgeon bases himself for this on imaging and peroperative vision. Unfortunately, this is not always sufficient and it is sometimes determined after surgery that the cutting edges are not free of tumor cells. Research has already shown that there is a significantly better survival when a margin of at least 1 mm is maintained between the macroscopic tumor and the cut surface. It is therefore important to remove the tumor as completely as possible without the risk of residual tissue and with a sufficiently wide margin.

The only method that can currently be used to determine during surgery if the tumor has been completely removed is to use "frozen sections". With a frozen section, the surgical piece is sent to the pathology department during the operation, where sections are taken from the edges. These are frozen in nitrogen and immediately viewed by a pathologist. If the cut edge is positive, this will be passed on to the surgeon who will take a wider resection if possible. Unfortunately, this method is time consuming and labor intensive. The evaluation of these cut edges on frozen section is not easy and requires a lot of experience. The percentage of false negative reviews for frozen section is not high, but it is true that it is not non-existent either. In addition, it is not possible to evaluate all cleavage surfaces peroperatively. This is currently happening for the distal pancreatic cutting edge and the bile duct cutting edge, but not, for example, for the posterior pancreatic surface and for the surface of the groove in which the superior mesenteric vein runs.

The use of peroperative imaging in the form of 18F-FDG PET-CT scan of the tumor would be a clear asset for this. This would not only be faster than frozen sections, but also provide a full 3-dimensional image of the extracted specimen, which may provide more insights than 2D frozen sections. The ultimate goal of this study is to bring the high resolution PET-CT system into the operating theater. For example, during the operation, in the operating theater itself, it could be determined where residual tumor tissue would be present and then performed a wider resection in order to avoid a positive margin status.

DETAILED DESCRIPTION:
This study will be conducted in patients undergoing surgery for pancreatic cancer removal. The aim of this study is to see whether all tumor tissue has been removed in this patient group during the removal of the tumor. This will be done with the help of a high resolution PET-CT (Positron Emission Tomography - Computer Tomography) system, developed by the Faculty of Engineering, UGent, and commercialized by Xeos (spin-off from Ghent University). This system is the compact (and transportable version) of the standard PET-CT and was initially developed for imaging small laboratory animals, typically mice, for which a particularly high resolution is required. In this study, the high-resolution PET-CT system will be used to evaluate the cutting edges after tumor resection. The goal is to evaluate the distance of the tumor cells from the cutting edges of the surgical piece.

The patient receives an intravenous injection of radiolabeled sugar (18F-FDG). 18F-FDG is the standard PET tracer for diagnostic PET-CT research. This standard dose will always be calculated according to the formula: 3.7 x body weight + 37 Mbq. The injection will be carried out by a trained "helper" under article 53.2 of the Royal Decree of 30/08/2001. This injection is always carried out under the responsibility of Dr. Kathia De Man or Dr. Bliede Van den Broeck as a recognized and licensed nuclear medicine doctor. The location of the injection will depend on the logistical possibilities of the day of operation. Due to the radioactive decay of the molecule, the optimal moment of injection of this radiolabeled sugar is best as short as possible before scanning the tumor. If possible, a "helper" will transport the radiolabelled sugar to the operating theater (OR) and the injection will be performed in the OR itself. If this option does not exist, the injection will be performed at the nuclear medicine department of UZ Gent, after which the injected patient will be immediately taken to the OR. Based on the natural decay of the radioactivity, the results of both injection times can be compared using the time of injection, injected dose and time of scan. The data collected during the study will allow to calculate post-hoc what the ideal dose of 18F-FDG is for this indication, i.e. the lowest possible dose for the patient, which can still be optimally measured by the scanner . The ALARA (as low as reasonably achievable) principle always applies.

The surgery to remove the pancreatic tumor follows the standard procedure. After removal, the surgical piece is first taken to the anatomopathology department. Frozen sections will be taken and analyzed directly for intake by tumor cells. Immediate feedback on this is given to the surgeon in the OR, as is done within the standard procedure. After taking the frozen sections, the rest of the specimen is taken to the "INFINITY" lab on the UZ Gent campus. Here a high-resolution PET-CT scan is performed on the surgical piece. After the PET-CT scan, the surgical piece is returned to the pathological anatomy department for further standard pathological evaluation. No information about the PET-CT results will be given to the surgeon during surgery so as not to interfere with the standard surgical procedure. The results of the high resolution PET-CT scan will be correlated post-hoc with the routine histopathological results of the tumor specimen, which is considered the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years)
* Signed informed consent
* Patient with a Pancreas Ca who is undergoing Whipple surgery
* Patient with ASA grade 1 to 3

Exclusion Criteria:

* Patient has ASA 4
* Patient under long-term use of anticoagulant therapy (except low dose aspirin)
* Patient has tumor invasion of blood vessels
* The patient undergoes a total pancreatectomy
* Patient undergoes a double derivation
* pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
marge assessment immediately after resection | marge assessment immediately performed results known after 3 weeks
  first PET imaging after resection for visiuallazation of the proximity of the leasion then frozen section of the cutting edge to astablising the same result and comparing the results from PET and frozen section.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD-PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, East-flanders, Belgium

IPD SHARING:
Plan to Share IPD: No